CLINICAL TRIAL: NCT00315328
Title: A Randomized Trial Comparing Patching Versus Atropine for Amblyopia in 7 to < 13 Year Olds
Brief Title: Trial Comparing Patching Versus Atropine for Amblyopia in 7 to < 13 Year Olds
Acronym: ATS9
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Ray Kraker, Director, PEDIG Coordinating Center, Jaeb Center for Health Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-119; 2U10EY011751 (NIH)
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Results first posted 2011-06-06 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Amblyopia
Keywords: Amblyopia; Atropine; Patching
MeSH Terms: conditions — Amblyopia | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patching (Active Comparator): Patching 2 hours per day plus near activities for one hour while patching (with increase to 4 hours per day for moderate amblyopes and >4 hours per day for severe amblyopes at 5 weeks if acuity not improved at least 5 letters)
  Interventions: Device: Patching; Procedure: Near activities
- Atropine (Active Comparator): Atropine 1% once each weekend day in the sound eye plus near activities for at least one hour every day (with increase to daily atropine at 5 weeks if acuity not improved by at least 5 letters)
  Interventions: Drug: Atropine; Procedure: Near activities

INTERVENTIONS:
Drug: Atropine — Atropine 1% each weekend day in the sound eye
  Arms: Atropine
Device: Patching — Patching 2 hours per day
  Other Names: Coverlet, 3M Opticlude, Ortopad®
  Arms: Patching
Procedure: Near activities — near visual activities for at least one hour per day

SUMMARY:
The purpose of this study is:

* To compare the effectiveness of weekend atropine plus near activities and daily patching plus near activities for moderate amblyopia (20/40 to 20/100) and severe amblyopia (20/125 to 20/400) in improving vision in the amblyopic eye of 7 to <13 year olds.
* To determine the maximum improvement in vision of the amblyopic eye with each treatment.
* To determine whether amblyopia is associated with structural abnormalities of optic nerve fiber layer.

DETAILED DESCRIPTION:
Although there is consensus that amblyopia can be treated effectively in young children, many eye care practitioners believe that treatment beyond a certain age is ineffective. Some clinicians have believed that a treatment response is unlikely after the age of 6 or 7 years, while others have considered age 9 or 10 years to be the upper age limit for successful treatment. The American Academy of Ophthalmology Preferred Practice Pattern for amblyopia recommends treatment up to age 10 years. The opinion that amblyopia treatment is ineffective in older children may have arisen because the age of 6 to 7 years is thought to be the end of the "critical period" for visual development in humans. This belief, however, was not based on adequate prospectively-collected data.

To address this issue of the response of amblyopia to treatment in children 7 years and older, the Pediatric Eye Disease Investigator Group (PEDIG) conducted a randomized trial of 507 patients (aged 7 to <18 years) with amblyopic eye visual acuity ranging from 20/40 to 20/400. Patients were provided with optimal optical correction and then randomized to a Treatment Group (2 to 6 hours per day of prescribed patching of the sound eye combined with near visual activities for all patients plus atropine one drop per day in the sound eye for 7 to <13 year olds) or an Optical Correction Group (optical correction alone). Patients whose amblyopic eye acuity improved 10 or more letters (2 lines) by 24 weeks were considered responders. In the 7 to <13 year olds (N=404), 53% of the Treatment Group were responders compared with 25% of the Optical Correction Group (P<0.001). In the 13 to <18 year olds (N=103), the responder rates were 25% and 23% respectively overall (adjusted P=0.22), but 47% and 20% respectively among patients not previously treated with patching and/or atropine for amblyopia (adjusted P=0.03). Most patients, including responders, were left with a residual visual acuity deficit.

The use of multiple modalities (patching, atropine, near visual activities) in the treatment regimen for the 7 to <13 year olds in this trial (ATS3) was an effort to maximize the therapeutic response. Patients age 13 years and older were prescribed patching but not atropine because of concern that the continual optical blur from the atropine could have a deleterious effect on their ability to drive and perform other activities. Prescribed patching was 2 to 6 hours a day to limit patch wear to non-school hours and because our prior studies of 3 to <7 year olds demonstrated that as little as two hours of patching a day (when combined with near visual activities) is as effective as a greater number of hours. Instructing patients to perform at least one hour of near activities while wearing the patch was based on the unproven clinical opinion that near activities can augment the effect of the occlusion therapy. A PEDIG pilot study suggested that near activities are beneficial and this question of benefit of near activities is currently being studied in another randomized clinical trial. Atropine placed in the sound eye once a day and two days a week has been demonstrated in younger children to be beneficial to the acuity of the amblyopic eye, presumably due to its cycloplegic effect of blurring vision in the sound eye especially at near fixation. In a study comparing daily and weekend atropine, daily atropine was not found to be superior.

The unanswered question from this completed clinical trial is whether prescribing patching or atropine alone could have produced a response similar to the combination therapy, or whether in this age group, one treatment is better than the other. A poll of PEDIG investigators at an investigator meeting on January 15, 2005 indicated that very few are following the treatment regimen used in the prior study (ATS3); rather, most are prescribing monotherapy-either patching or atropine-as the initial treatment for amblyopia in the 7 to <13 year age range. Thus, a trial comparing atropine and patching as amblyopia treatments in 7 to <13 year olds is needed.

The study has been designed as a simple trial that, other than the type of amblyopia therapy being determined through the randomization process, approximates standard clinical practice. The two treatment regimes are: 1) Atropine 1% once each weekend day in the sound eye plus near activities for at least one hour every day without the aid of reading glasses (with increase to daily atropine at 5 weeks if acuity not improved by at least 5 letters) and 2) Patching 2 hours per day plus near activities for one hour while patching (with increase to 4 hours per day for moderate amblyopes and > 4 hours per day for severe amblyopes at 5 weeks if acuity not improved by at least 5 letters).

Optional Ancillary Study As part of the optic nerve imaging ancillary study, retinal nerve fiber layer imaging using optical coherence tomography will be performed on some patients. This will be optional for patients at participating sites. The procedure is not part of standard care. The subject's pupils will need to be dilated, if not already dilated as part of the exam. Testing of both eyes can be completed in about 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 7 to 12 years old (inclusive)
* Amblyopia associated with strabismus, anisometropia, or both
* Visual acuity in the amblyopic eye 19 to 71 letters on Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS©) (20/40 to 20/400 inclusive)
* Visual acuity in the sound eye 79 letters or better on E-ETDRS© (20/25 or better)
* Interocular difference >=15 letters (3 lines)
* Spectacles, if needed, worn for at least 16 weeks or visual acuity documented to be stable

Inclusion Criteria for Optional Ancillary Study:

* Enrolled into the main study
* Refractive error in both eyes between -0.25 and +5.00D, inclusive (to avoid the need to adjust for refractive error)
* Birth weight >1500 grams
* No history of Central Nervous System (CNS) disease (e.g. intraventricular hemorrhage (IVH), periventricular leukomalacia (PVL), meningitis, developmental abnormalities of the brain, hydrocephalus, cerebral palsy, hypoxic ischemic encephalopathy

Exclusion Criteria:

* Amblyopia treatment (other than spectacles) in the last 6 months
* Myopia (more than -0.25D spherical equivalent) in either eye

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 233 (Actual)
Dates: Start 2005-08; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W. Hertle, M.D., Study Chair — University of Pittsburgh; Mitchell M. Scheiman, O.D., Study Chair — Pennsylvania College of Optometry
Locations (2):
- United States (2):
  - Pennsylvania College of Optometry, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Repka MX, Kraker RT, Beck RW, Birch E, Cotter SA, Holmes JM, Hertle RW, Hoover DL, Klimek DL, Marsh-Tootle W, Scheiman MM, Suh DW, Weakley DR; Pediatric Eye Disease Investigator Group. Treatment of severe amblyopia with weekend atropine: results from 2 randomized clinical trials. J AAPOS. 2009 Jun;13(3):258-63. doi: 10.1016/j.jaapos.2009.03.002. PMID 19541265
- [Background] Repka MX, Kraker RT, Tamkins SM, Suh DW, Sala NA, Beck RW; Pediatric Eye Disease Investigator Group. Retinal nerve fiber layer thickness in amblyopic eyes. Am J Ophthalmol. 2009 Jul;148(1):143-7. doi: 10.1016/j.ajo.2009.01.015. Epub 2009 Mar 27. PMID 19327749
- [Background] Pediatric Eye Disease Investigator Group. Pharmacological plus optical penalization treatment for amblyopia: results of a randomized trial. Arch Ophthalmol. 2009 Jan;127(1):22-30. doi: 10.1001/archophthalmol.2008.520. PMID 19139333
- [Background] Felius J, Chandler DL, Holmes JM, Chu RH, Cole SR, Hill M, Huang K, Kulp MT, Lazar EL, Matta NS, Melia M, Wallace DK; Pediatric Eye Disease Investigator Group. Evaluating the burden of amblyopia treatment from the parent and child's perspective. J AAPOS. 2010 Oct;14(5):389-95. doi: 10.1016/j.jaapos.2010.07.009. PMID 21035063
- [Result] Scheiman MM, Hertle RW, Kraker RT, Beck RW, Birch EE, Felius J, Holmes JM, Kundart J, Morrison DG, Repka MX, Tamkins SM; Pediatric Eye Disease Investigator Group. Patching vs atropine to treat amblyopia in children aged 7 to 12 years: a randomized trial. Arch Ophthalmol. 2008 Dec;126(12):1634-42. doi: 10.1001/archophthalmol.2008.107. PMID 19064841
- [Derived] Wallace DK, Lazar EL, Melia M, Birch EE, Holmes JM, Hopkins KB, Kraker RT, Kulp MT, Pang Y, Repka MX, Tamkins SM, Weise KK; Pediatric Eye Disease Investigator Group. Stereoacuity in children with anisometropic amblyopia. J AAPOS. 2011 Oct;15(5):455-61. doi: 10.1016/j.jaapos.2011.06.007. PMID 22108357
- [Derived] Repka M, Simons K, Kraker R; Pediatric Eye Disease Investigator Group. Laterality of amblyopia. Am J Ophthalmol. 2010 Aug;150(2):270-4. doi: 10.1016/j.ajo.2010.01.040. Epub 2010 May 8. PMID 20451898
- See also: PubMed Abstract — https://www.ncbi.nlm.nih.gov/pubmed/19064841
- See also: PubMed Central HHS Public Access - Full Text — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2846774/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2005 and July 2007, 233 subjects were randomized at 39 certified sites (193 with moderate amblyopia 20/40 to 20/100 in a primary cohort, and an additional 40 with severe amblyopia 20/125 to 20/400 that were followed as a secondary cohort).
Pre-assignment Details: Subjects must have been wearing optimal spectacle correction for a minimum of 16 weeks or until stability of visual acuity was documented (no improvement in amblyopic eye visual acuity at 2 consecutive visits at least 4 weeks apart) before enrollment and randomization.
Groups:
- Patching-Moderate Amblyopia: Patching 2 hours per day plus near activities for one hour while patching among patients with moderate amblyopia (20/40 to 20/100)
- Atropine-Moderate Amblyopia: Atropine 1% once each weekend day in the sound eye plus near activities for at least one hour every day among patients with moderate amblyopia (20/40 to 20/100).
- Patching-Severe Amblyopia: Patching 2 hours per day plus near activities for one hour while patching among patients with severe amblyopia (20/125 to 20/400)
- Atropine-Severe Amblyopia: Atropine 1% once each weekend day in the sound eye plus near activities for at least one hour every day among patients with severe amblyopia (20/125 to 20/400).
Period: Overall Study
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Started | 98 (Includes subjects with moderate amblyopia only (20/40 to 20/100 at baseline)) | 95 (Includes subjects with moderate amblyopia only (20/40 to 20/100 at baseline)) | 18 (Includes subjects with severe amblyopia only (20/125 to 20/400 at baseline)) | 22 (Includes subjects with severe amblyopia only (20/125 to 20/400 at baseline))
5 Week Visit | 91 | 89 | 17 | 19
Completed | 84 (Completed defined as completing 17 week primary outcome exam) | 88 (Completed defined as completing 17 week primary outcome exam) | 13 (Completed defined as completing 17 week primary outcome exam) | 20 (Completed defined as completing 17 week primary outcome exam)
Not Completed | 14 | 7 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia | Total
Number analyzed (Participants) | 98 | 95 | 18 | 22 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at enrollment
  years | 8.9 (1.5) | 9.1 (1.6) | 9.5 (1.5) | 9.2 (1.8) | 9.0 (1.6)
Age, Customized [Number; unit: participants] — Age at enrollment
  participants
    7 to <8 years | 35 | 28 | 6 | 9 | 78
    8 to <9 years | 24 | 26 | 0 | 4 | 54
    9 to <10 years | 17 | 16 | 5 | 3 | 41
    10 to <11 years | 8 | 10 | 4 | 2 | 24
    11 to <12 years | 8 | 7 | 2 | 1 | 18
    12 to <13 years | 6 | 8 | 1 | 3 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 54 | 4 | 12 | 118
  Male | 50 | 41 | 14 | 10 | 115
Race/Ethnicity, Customized [Number; unit: participants]
  White | 68 | 56 | 16 | 18 | 158
  African-American | 8 | 11 | 2 | 1 | 22
  Hispanic or Latino | 20 | 23 | 0 | 3 | 46
  Asian | 0 | 1 | 0 | 0 | 1
  More than one race | 1 | 2 | 0 | 0 | 3
  Not reported | 1 | 2 | 0 | 0 | 3
Cause of Amblyopia [Number; unit: participants]
  Strabismus | 28 | 33 | 4 | 4 | 69
  Anisometropia | 46 | 31 | 6 | 9 | 92
  Strabismus and anisometropia | 24 | 31 | 8 | 9 | 72
Distance Visual Acuity in Amblyopic Eye [Number; unit: participants] — Visual acuity was measured in each eye using the electronic early treatment diabetic retinopathy study (E-ETDRS) method which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
  participants
    20/400 (18 to 22 letters) (worse) | 0 | 0 | 0 | 1 | 1
    20/320 (23 to 27 letters) | 0 | 0 | 0 | 1 | 1
    20/250 (28 to 32 letters) | 0 | 0 | 2 | 4 | 6
    20/200 (33 to 37 letters) | 0 | 0 | 8 | 3 | 11
    20/160 (38 to 42 letters) | 0 | 0 | 5 | 4 | 9
    20/125 (43 to 47 letters) | 0 | 0 | 3 | 9 | 12
    20/100 (48 to 52 letters) | 6 | 13 | 0 | 0 | 19
    20/80 (53 to 57 letters) | 15 | 13 | 0 | 0 | 28
    20/63 (58 to 62 letters) | 24 | 22 | 0 | 0 | 46
    20/50 (63 to 67 letters) | 33 | 28 | 0 | 0 | 61
    20/40 (68 to 72 letters) (best) | 20 | 19 | 0 | 0 | 39
Distance Visual Acuity in Fellow Eye [Number; unit: participants] — Visual acuity was measured in each eye using the electronic early treatment diabetic retinopathy study (E-ETDRS) method which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
  participants
    20/32 (73 to 77 letters) (worse) | 0 | 0 | 0 | 0 | 0
    20/25 (78 to 82 letters) | 17 | 20 | 1 | 6 | 44
    20/20 (83 to 87 letters) | 43 | 47 | 8 | 5 | 103
    20/16 (88 to 92 letters) | 36 | 26 | 9 | 11 | 82
    20/12 (93 to 97 letters) (best) | 2 | 2 | 0 | 0 | 4
Prior Treatment for Amblyopia at Enrollment [Number; unit: participants]
  None | 71 | 68 | 13 | 18 | 170
  Patching | 16 | 16 | 2 | 3 | 37
  Atropine | 2 | 0 | 1 | 0 | 3
  Patching and atropine | 9 | 11 | 2 | 1 | 23
Refractive Error in Amblyopic Eye (spherical equivalent) [Number; unit: participants] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. Spherical equivalent is defined as the sphere plus 1/2 the cylinder.
  participants
    < 0 Diopters (D) | 2 | 2 | 0 | 0 | 4
    0 to < +1.00D | 8 | 10 | 1 | 1 | 20
    +1.00 to < +2.00D | 13 | 6 | 2 | 2 | 23
    +2.00 to < +3.00D | 10 | 8 | 1 | 3 | 22
    +3.00 to < +4.00D | 23 | 16 | 2 | 4 | 45
    >= +4.00D | 42 | 53 | 12 | 12 | 119
Refractive Error in Fellow Eye (spherical equivalent) [Number; unit: participants] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. Spherical equivalent is defined as the sphere plus 1/2 the cylinder.
  participants
    < 0 Diopters (D) | 1 | 2 | 0 | 0 | 3
    0 to < +1.00D | 32 | 29 | 4 | 9 | 74
    +1.00 to < +2.00D | 33 | 17 | 8 | 5 | 63
    +2.00 to < +3.00D | 13 | 9 | 1 | 2 | 25
    +3.00 to < +4.00D | 7 | 6 | 2 | 2 | 17
    >= +4.00D | 12 | 32 | 3 | 4 | 51
Distance Visual Acuity in Amblyopic Eye [Mean (Standard Deviation); unit: ETDRS letter score] — Visual acuity was measured in each eye using the electronic early treatment diabetic retinopathy study (E-ETDRS) method which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
  ETDRS letter score | 62.4 (5.7) | 61.7 (6.6) | 37.5 (5.0) | 37.5 (7.5) | 57.9 (11.1)
Distance Visual Acuity in Fellow Eye [Mean (Standard Deviation); unit: ETDRS letter score] — Visual acuity was measured in each eye using the electronic early treatment diabetic retinopathy study (E-ETDRS) method which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
  ETDRS letter score | 86.0 (3.6) | 85.7 (3.4) | 87.0 (3.5) | 85.5 (4.0) | 85.9 (3.6)
Intereye Acuity Difference [Mean (Standard Deviation); unit: ETDRS letter score] — Visual acuity was measured in each eye using the electronic early treatment diabetic retinopathy study (E-ETDRS) method which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. Intereye difference defined as the difference between ETDRS letter scores (amblyopic eye minus sound eye).
  ETDRS letter score | 23.5 (6.8) | 24.0 (7.0) | 49.5 (5.5) | 47.5 (9.5) | 28.0 (11.7)
Refractive Error in Amblyopic Eye (spherical equivalent [Mean (Standard Deviation); unit: diopter] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. Spherical equivalent is defined as the sphere plus 1/2 the cylinder.
  diopter | 3.57 (2.07) | 4.10 (2.19) | 4.97 (2.50) | 4.18 (1.99) | 3.95 (2.16)
Refractive Error in Fellow Eye (spherical equivalent) [Mean (Standard Deviation); unit: diopter] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. Spherical equivalent is defined as the sphere plus 1/2 the cylinder.
  diopter | 1.84 (1.74) | 2.56 (2.22) | 2.12 (1.76) | 1.98 (2.11) | 2.17 (2.00)

OUTCOME MEASURES:

1. Secondary Outcome: Stereoacuity Measured by the Randot Preschool Test at 17 or 19 Weeks- Participants With All Causes of Moderate Amblyopia
Description: The Randot Preschool Stereotest measures stereopsis from 800 to 40 seconds of arc on patients as young as 2 years of age. This Stereotest is designed as a matching game in which the patient matches pictures in a test booklet wearing special glasses. A subject can fail the pretest (not see any pictures) or can score >800 (the worst), 800, 400, 200, 100, 60, or 40 (the best) seconds of arc. If two shapes are identified correctly the patient progresses to the next lower stereoacuity level. A failed test occurs when the patient cannot identify any shapes.
Time Frame: 17 or 19 weeks
Measure: Number; unit: Participants
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 0 | 0
Participants
  Failed black & white shape identification pretest | 1 | 4 |  |
  >800 arcsec (worse) | 26 | 34 |  |
  800 arcsec | 9 | 3 |  |
  400 arcsec | 9 | 14 |  |
  200 arcsec | 10 | 10 |  |
  100 arcsec | 9 | 12 |  |
  60 arcsec | 7 | 2 |  |
  40 arcsec (best) | 13 | 9 |  |
Statistical Analysis 1: Comparison: Patching-Moderate Amblyopia vs Atropine-Moderate Amblyopia; Wilcoxon rank sum tests were used to assess treatment group differences in the change in Randot Preschool stereoacuity levels ( from baseline to the outcome examination); Test type: Superiority or Other; p = 0.96, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Stereoacuity Measured by the Randot Preschool Test at 17 or 19 Weeks- Anisometropic Participants With Moderate Amblyopia Only
Description: as for outcome 1
Time Frame: 17 or 19 weeks
Measure: Number; unit: Participants
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 42 | 28 | 0 | 0
Participants
  Failed black & white shape identification pretest | 0 | 0 |  |
  >800 arcsec (worse) | 5 | 6 |  |
  800 arcsec | 3 | 1 |  |
  400 arcsec | 5 | 4 |  |
  200 arcsec | 7 | 4 |  |
  100 arcsec | 9 | 8 |  |
  60 arcsec | 6 | 0 |  |
  40 arcsec (best) | 7 | 5 |  |
Statistical Analysis 1: Comparison: Patching-Moderate Amblyopia vs Atropine-Moderate Amblyopia; Wilcoxon rank sum tests used to assess treatment group differences in change in Randot Preschool stereoacuity levels ( from baseline to the outcome examination) among those with anisometropia only; Test type: Superiority or Other; p = 0.78, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Stereoacuity Measured by the Randot Preschool Test at 17 or 19 Weeks- Participants With Moderate Amblyopia From Strabismus Only or Combined Mechanism
Description: as for outcome 1
Time Frame: 17 or 19 weeks
Measure: Number; unit: Participants
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 42 | 60 | 0 | 0
Participants
  Failed black & white shape identification pretest | 1 | 4 |  |
  >800 arcsec (worse) | 21 | 28 |  |
  800 arcsec | 6 | 2 |  |
  400 arcsec | 4 | 10 |  |
  200 arcsec | 3 | 6 |  |
  100 arcsec | 0 | 4 |  |
  60 arcsec | 1 | 2 |  |
  40 arcsec (best) | 6 | 4 |  |
Statistical Analysis 1: Comparison: Patching-Moderate Amblyopia vs Atropine-Moderate Amblyopia; Wilcoxon rank sum tests were used to assess treatment group differences in the change in Randot Preschool stereoacuity levels ( from baseline to the outcome examination) among patients with strabismus or combined mechanism only; Test type: Superiority or Other; p = 0.99, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Stereoacuity Measured by the Randot Preschool Test at 17 or 19 Weeks- Participants With All Causes of Moderate Amblyopia
Description: Stereoacuity is scored as seconds of arc with values of: <800, 800, 400, 200, 100, 60, 40. The lower the arc second value, the better the score (i.e. 40 arc sec is best stereoacuity; <800 is the worst). A change score was defined as the difference between baseline and outcome in score level (i.e. moving from 800 at baseline to 400 at outcome is one level change, moving from 800 to 200 is two levels, etc.) change in levels was categorized as "within one level" meaning change was -1, 0, or +1.
Time Frame: 17 or 19 weeks
Measure: Number; unit: Participants
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 0 | 0
Participants
  >= 2 levels worse | 4 | 9 |  |
  Within 1 level | 57 | 54 |  |
  >= 2 levels better | 17 | 18 |  |
Statistical Analysis 1: Comparison: Atropine-Moderate Amblyopia; To evaluate WITHIN each treatment group whether stereoacuity changed from baseline to outcome a Wilcoxon sign-rank test was performed to evaluate whether the distribution of change from baseline was zero; Test type: Superiority or Other; p = .04, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Patching-Moderate Amblyopia; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Amblyopia Treatment Index - Social Stigma (Moderate Amblyopia Only)
Description: Questionnaire scores on the Social Stigma subscale of the Amblyopia Treatment Index. Questions were evaluated on a likert type scale as strongly agree (5) to strongly disagree (1), with a higher number indicating worse response.
Time Frame: 17 weeks
Population: Number of subjects who completed the 17wk amblyopia treatment index questionnaire evaluating the impact of treatment on the child and family.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 66 | 64 | 0 | 0
Units on a scale | 2.37 (0.75) | 1.91 (0.75) |  |
Statistical Analysis 1: Comparison: Patching-Moderate Amblyopia; Wilcoxon rank sum tests were used to assess treatment group differences in the parent questionnaire subscale scores at 17 weeks - Social Stigma subscale; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney); Positive mean favors atropine group

6. Secondary Outcome: Amblyopia Treatment Index - Compliance (Moderate Amblyopia Only)
Description: Questionnaire scores on the compliance subscale of the Amblyopia Treatment Index. Questions were evaluated on a likert type scale as strongly agree (5) to strongly disagree (1), with a higher number indicating worse response.
Time Frame: 17 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 66 | 64 | 0 | 0
Units on a scale | 2.59 (0.93) | 2.03 (0.82) |  |
Statistical Analysis 1: Comparison: Patching-Moderate Amblyopia vs Atropine-Moderate Amblyopia; Wilcoxon rank sum tests were used to assess treatment group differences in the parent questionnaire subscale scores at 17 weeks - Compliance subscale; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney); Positive mean favors atropine group

7. Secondary Outcome: Amblyopia Treatment Index - Adverse Effects Scale (Moderate Amblyopia Only)
Description: Questionnaire scores on the adverse events subscale of the Amblyopia Treatment Index. Questions were evaluated on a likert type scale as strongly agree (5) to strongly disagree (1), with a higher number indicating worse response.
Time Frame: 17 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 66 | 64 | 0 | 0
Units on a scale | 2.28 (0.68) | 2.22 (0.80) |  |
Statistical Analysis 1: Comparison: Patching-Moderate Amblyopia vs Atropine-Moderate Amblyopia; Wilcoxon rank sum tests were used to assess treatment group differences in the parent questionnaire subscale scores at 17 weeks - Adverse events subscale; Test type: Superiority or Other; p = 0.70, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Distribution of Visual Acuity in the Amblyopic Eye at 17 Weeks
Description: Visual acuity was measured in each eye using the electronic early treatment diabetic retinopathy study (E-ETDRS) method which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
Time Frame: 17 weeks
Population: Primary analysis includes only patients who completed the 17 week exam between 13 and 26 weeks following randomization. No imputation was done if missed exam; analysis followed the intent to treat principle.
Measure: Number; unit: participants
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 13 | 20
participants
  20/400 (18 to 22 letters) (worse) | 0 | 0 | 0 | 0
  20/320 (23 to 27 letters) | 0 | 0 | 0 | 1
  20/250 (28 to 32 letters) | 0 | 0 | 0 | 3
  20/200 (33 to 37 letters) | 0 | 0 | 3 | 3
  20/160 (38 to 42 letters) | 1 | 0 | 1 | 3
  20/125 (43 to 47 letters) | 0 | 1 | 4 | 2
  20/100 (48 to 52 letters) | 3 | 4 | 1 | 2
  20/80 (53 to 57 letters) | 3 | 6 | 4 | 3
  20/63 (58 to 62 letters) | 5 | 12 | 0 | 1
  20/50 (63 to 67 letters) | 13 | 14 | 0 | 1
  20/40 (68 to 72 letters) | 20 | 15 | 0 | 0
  20/32 (73 to 77 letters) | 19 | 21 | 0 | 0
  20/25 (78 to 82 letters) | 14 | 10 | 0 | 1
  20/20 (83 to 87 letters) | 6 | 4 | 0 | 0
  20/16 (88 to 92 letters) (best) | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Patching-Moderate Amblyopia vs Atropine-Moderate Amblyopia; 95% confidence interval constructed on the treatment group difference in proportion with amblyopic eye visual acuity 20/25 or better at 17 weeks; Test type: Superiority or Other; Mean Difference (Net) = 0.07, 95% CI [-0.03 to 0.17]

9. Primary Outcome: Mean Visual Acuity in the Amblyopic Eye at 17 Weeks
Description: as for outcome 8
Time Frame: 17 weeks
Measure: Mean (Standard Deviation); unit: ETDRS letter score
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 13 | 20
ETDRS letter score | 71.0 (8.9) | 69.2 (9.2) | 46.0 (6.0) | 45.0 (14.0)

10. Primary Outcome: Distribution of Change in Visual Acuity in the Amblyopic Eye From Baseline to 17 Weeks
Description: Visual acuity was measured at baseline and 17 weeks in each eye using the electronic early treatment diabetic retinopathy study (E-ETDRS) method which resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. A difference between the scores at baseline and 17 weeks was calculated.
  A positive difference indicates acuity was better at 17 weeks than at baseline; a negative difference indicates acuity was worse at 17 weeks.
Time Frame: Baseline to 17 weeks
Measure: Number; unit: participants
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 13 | 20
participants
  >=15 letters worse | 1 | 0 | 0 | 0
  10 to 14 letters worse | 0 | 2 | 0 | 0
  5 to 9 letters worse | 0 | 3 | 0 | 2
  +/- 4 letters | 23 | 22 | 2 | 6
  5 to 9 letters better | 22 | 26 | 4 | 4
  10 to 14 letters better | 17 | 20 | 2 | 3
  >=15 letters better | 21 | 15 | 5 | 5
Statistical Analysis 1: Comparison: Patching-Moderate Amblyopia vs Atropine-Moderate Amblyopia; 95% confidence interval constructed on the treatment group difference of the proportion improving 15 or more letters from baseline to 17 weeks; Test type: Superiority or Other; Mean Difference (Net) = 0.08, 95% CI [-0.02 to 0.18]

11. Primary Outcome: Mean Change in Visual Acuity in the Amblyopic Eye From Baseline to 17 Weeks
Description: as for outcome 10
Time Frame: Baseline to 17 weeks
Measure: Mean (Standard Deviation); unit: ETDRS letter score
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 13 | 20
ETDRS letter score | 8.6 (7.8) | 7.6 (7.5) | 9.0 (6.5) | 7.5 (10.5)
Statistical Analysis 1: Comparison: Patching-Moderate Amblyopia vs Atropine-Moderate Amblyopia; The trial was designed to evaluate whether patching and atropine are equivalent treatments for amblyopia in children 7 to 12 years old. The sample size was computed based on a standard deviation of 17-week visual acuity scores of 10 letters, correlation between outcome and baseline visual acuity scores of 0.30 and 10% loss to follow up; Test type: Non-Inferiority or Equivalence — Treatment equivalence was to be declared if the ends of the 2 1-sided 95% confidence intervals constructed on the difference between adjusted mean visual acuity scores were completely contained within the designated equivalence interval of +/- 5 letters; ANCOVA; Mean Difference (Net) = 1.2, 95% CI [-0.7 to 3.1]

12. Secondary Outcome: Distribution of Visual Acuity in the Fellow Eye at 17 Weeks
Description: as for outcome 8
Time Frame: 17 weeks
Measure: Number; unit: participants
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 13 | 20
participants
  20/50 (63 to 67 letters) (worse) | 0 | 0 | 0 | 0
  20/40 (68 to 72 letters) | 0 | 0 | 0 | 1
  20/32 (73 to 77 letters) | 2 | 4 | 0 | 1
  20/25 (78 to 82 letters) | 5 | 12 | 1 | 2
  20/20 (83 to 87 letters) | 31 | 42 | 4 | 4
  20/16 (88 to 92 letters) | 42 | 29 | 5 | 11
  20/12 (93 to 97 letters) (best) | 4 | 1 | 3 | 1

13. Secondary Outcome: Mean Visual Acuity in the Fellow Eye at 17 Weeks
Description: as for outcome 8
Time Frame: 17 weeks
Measure: Mean (Standard Deviation); unit: ETDRS letter score
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 13 | 20
ETDRS letter score | 87.3 (3.8) | 85.8 (3.9) | 88.5 (5.0) | 86.5 (6.5)

14. Secondary Outcome: Distribution of Change in Visual Acuity in the Fellow Eye From Baseline to 17 Weeks
Description: as for outcome 10
Time Frame: Baseline to 17 weeks
Measure: Number; unit: participants
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 13 | 20
participants
  >=10 letters worse | 0 | 0 | 0 | 1
  5 to 9 letters worse | 4 | 7 | 1 | 2
  +/- 4 letters | 69 | 72 | 8 | 11
  5 to 9 letters better | 11 | 9 | 4 | 4
  >=10 letters better | 0 | 0 | 0 | 2
Statistical Analysis 1: Comparison: Patching-Moderate Amblyopia vs Atropine-Moderate Amblyopia; 95% confidence interval constructed on the treatment group difference of mean change in fellow eye visual acuity from baseline to 17 weeks, adjusted for baseline fellow eye visual acuity; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 1.3, 95% CI 2-sided [0.4 to 2.2]

15. Secondary Outcome: Mean Change in Visual Acuity in the Fellow Eye From Baseline to 17 Weeks
Description: as for outcome 10
Time Frame: Baseline to 17 weeks
Measure: Mean (Standard Deviation); unit: ETDRS letter score
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Number analyzed (Participants) | 84 | 88 | 13 | 20
ETDRS letter score | 1.5 (3.1) | 0.3 (3.5) | 1.0 (3.0) | 1.0 (5.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the 17 week outcome visit.
Arm/Group | Patching-Moderate Amblyopia | Atropine-Moderate Amblyopia | Patching-Severe Amblyopia | Atropine-Severe Amblyopia
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/95 | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 0/98 | 14/95 | 0/18 | 5/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patching-Moderate Amblyopia (N=98) | Atropine-Moderate Amblyopia (N=95) | Patching-Severe Amblyopia (N=18) | Atropine-Severe Amblyopia (N=22)
Light sensitivity (Eye disorders) | 0 | 14 | 0 | 3
Systemic (General disorders) | 0 | 0 | 0 | 2 — Systemic side effects were reported by 2 subjects using atropine - 1 reported irritability, and another reported urinary urgency, dry mouth, and excessive thirst.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No